CLINICAL TRIAL: NCT04544293
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial of Once-daily Inhaled Molgramostim Nebulizer Solution in Adult Subjects With Autoimmune Pulmonary Alveolar Proteinosis (aPAP)
Brief Title: Clinical Trial of Inhaled Molgramostim Nebulizer Solution in Autoimmune Pulmonary Alveolar Proteinosis (aPAP)
Acronym: IMPALA-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Savara Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAV006-05; 2020-001263-85 (EudraCT Number)
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Autoimmune Pulmonary Alveolar Proteinosis
Keywords: aPAP
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis, Acquired | interventions — molgramostim; Colony-Stimulating Factors; regramostim

STUDY DESIGN:
Intervention Model Description: Subject will be randomized 1:1 to treatment with inhaled molgramostim or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Molgramostim (Experimental): Double-blind treatment with molgramostim nebulizer solution 300 µg once daily (Mol OD) for 48 weeks
  Interventions: Drug: Molgramostim
- Placebo (Placebo Comparator): Double-blind treatment with placebo (PBO) nebulizer solution once daily for 48 weeks
  Interventions: Drug: Placebo
- Molgramostim Open-label Extension (Experimental): Open-label treatment with molgramostim nebulizer solution 300 µg once daily (Mol OD) for 96 weeks
  Interventions: Drug: Molgramostim Open-label

INTERVENTIONS:
Drug: Molgramostim — Molgramostim 300 µg nebulizer solution
  Other Names: Recombinant human granulocyte-macrophage colony stimulating factor (rhGM-CSF)
  Arms: Molgramostim
Drug: Placebo — Matching placebo nebulizer solution
  Other Names: Placebo nebulizer
  Arms: Placebo
Drug: Molgramostim Open-label — Molgramostim 300 µg nebulizer solution
  Other Names: Recombinant human granulocyte-macrophage colony stimulating factor (rhGM-CSF)
  Arms: Molgramostim Open-label Extension

SUMMARY:
160 subjects with autoimmune pulmonary alveolar proteinosis (aPAP) will be randomized to receive once daily treatment with inhaled molgramostim (MOL) or placebo (PBO) for 48 weeks. Subjects completing the 48-week placebo-controlled period will receive open-label treatment with once daily inhaled molgramostim for 96 weeks.

DETAILED DESCRIPTION:
This is an interventional, randomized, double-blind, 2-arm, parallel groups, placebo-controlled, multi-center, phase 3 trial in adult subjects who are diagnosed with aPAP.

An aPAP diagnosis should be confirmed by a Granulocyte-macrophage colony stimulating factor (GM-CSF) auto-antibody test result, and history of PAP based on either high resolution computed tomography, lung biopsy, or bronchoalveolar lavage cytology, should be available.

The trial consists of a 6-week screening period, a 48-week randomized, double-blind treatment period, a 96-week open-label treatment period, and a conditional 4-week safety follow-up period. The maximum treatment duration will be 145 weeks and the maximum trial duration will be 156 weeks. During the trial, whole lung lavage will be allowed as rescue treatment in case of worsening of aPAP.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be ≥18 years of age, at the time of signing the informed consent (≥20 in Japan).
2. A serum anti-GM-CSF autoantibody test result confirming autoimmune PAP.
3. History of PAP, based on examination of a lung biopsy, bronchoalveolar lavage (BAL) cytology, or a high-resolution computed tomogram (HRCT) of the chest.
4. A diffusing capacity for carbon monoxide of 70% predicted or lower adjusted for hemoglobin (%DLCOadj) at the screening and baseline visits.
5. Change in %DLCO adj of <15% points during the screening period.
6. Demonstrated functional impairment in the treadmill exercise test (defined as a peak metabolic equivalent (MET) ≤8).
7. Willing and able to come off supplemental oxygen use prior to and during the treadmill exercise test, the DLCO assessment, and the arterial blood gas sampling.
8. Resting oxygen saturation (SpO2) >85% during 15 minutes without use of supplemental oxygen at the screening visits.
9. Male or female
10. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

    1. Male subjects: Males agreeing to use condoms during and until 30 days after last dose of trial treatment, or males having a female partner who is using adequate contraception as described below.
    2. Female subjects: Females who have been post-menopausal for >1 year, or females of childbearing potential after a confirmed menstrual period using a highly efficient method of contraception (i.e. a method with <1% failure rate such as combined hormonal contraception, progesterone-only hormonal contraception, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner, sexual abstinence*), during and until 30 days after last dose of trial treatment. Females of childbearing potential must have a negative serum pregnancy test at the screening visits, and a negative urine pregnancy test at Baseline visit (Visit 3) and must not be lactating.
11. Capable of giving signed informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
12. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures specified in the protocol as judged by the Investigator.

Exclusion Criteria:

1. Diagnosis of hereditary or secondary PAP, or a metabolic disorder of surfactant production.
2. Whole lung lavage (WLL) performed within 3 months prior to baseline.
3. Requirement for WLL at screening or baseline.
4. GM-CSF treatment within 6 months prior to baseline.
5. Treatment with rituximab within 6 months prior to baseline.
6. Treatment with plasmapheresis within 6 weeks prior to baseline.
7. Treatment with any investigational medicinal product within 5 half-lives or 3 months (whichever is longer) prior to baseline.
8. Previously randomized in this trial.
9. History of allergic reactions to GM-CSF or any of the excipients in the nebulizer solution.
10. Inflammatory or autoimmune disease of a severity that necessitates significant (e.g. more than 10 mg/day systemic prednisolone) immunosuppression.
11. Previous experience of severe and unexplained side-effects during aerosol delivery of any kind of medicinal product.
12. History of, or present, myeloproliferative disease or leukemia.
13. Apparent pre-existing concurrent pulmonary fibrosis.
14. Acute or unstable cardiac or pulmonary disease that may be aggravated by exercise.
15. Known active infection (viral, bacterial, fungal, or mycobacterial) that may affect the efficacy evaluation in the trial.
16. Physical disability or other condition that precludes safe and adequate exercise testing.
17. Any other serious medical condition which in the opinion of the Investigator would make the subject unsuitable for the trial.
18. Pregnant, planning to become pregnant during the trial, or breastfeeding woman. For France only: including as further defined by French Health Code L-1121-5.
19. For France only: Any subject considered to be "vulnerable" on account of, e.g., mental or physical disability, socio-economic situation, or subjects deprived of their liberty. For France only: including as further defined by French Health Code L1121-8-1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2027-05-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Trapnell, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (54):
- United States (16):
  - University Of Arkansas For Medical Services, Little Rock, Arkansas
  - UCLA David Geffen School of Medicine, Los Angeles, California
  - National Jewish Health, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - University of Florida Health, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Loyola University, Maywood, Illinois
  - University of Maryland Medical Center, Baltimore, Maryland
  - Washington University in St. Louis, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Wake Med Health & Hospital, Raleigh, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania Perelman School of Medicine - Pulmonology, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Westmead Hospital, Westmead, New South Wales
- Belgium (2):
  - Hôpital Erasme, Brussels, Brussels Capital
  - UZ Leuven - Campus Gasthuisberg - Pneumologie, Leuven, Vlaams Brabant
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - St Joseph's Healthcare Hamilton Research, Hamilton, Ontario
  - University Institute of Cardiology and Respirology of Quebec, Québec
- France (2):
  - Hôpital Louis Pradel, Bron, Auvergne-Rhône-Alpes
  - CHU Pontchaillou, Rennes, Brittany Region
- Germany (3):
  - Thoraxklinik Heidelberg gGmbH am Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Asklepios Fachkliniken Muenchen-Gauting, Muenchen-Gauting, Bavaria
  - Ruhrlandklinik Westdeutsches Lungenzentrum, Essen, North Rhine-Westphalia
- Attikon University Hospital, Athens, Greece
- St. Vincent's University Hospital, Dublin, Ireland
- Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy
- Japan (9):
  - Hokkaido University Hospital, Sapporo, Hokkaidô
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama, Kanagawa
  - Tohoku University Hospital - Respiratory Tract Medicine, Sendai, Miyagi
  - National Hospital Organization Kinki-Chuo Chest medical Center, Sakai, Osaka
  - Kyorin University Hospital, Mitaka, Tokyo
  - Chiba University Hospital - Respiratory Medicine, Chiba
  - Kumamoto University Hospital, Kumamoto
  - Aichi Medical University Hospital, Nagakute
  - Saitama Red Cross Hospital, Saitama
- St Antonius Hospital, Nieuwegein, Utrecht, Netherlands
- Instytut Gruzlicy i Chorob Pluc, Warsaw, Masovian Voivodeship, Poland
- Portugal (2):
  - Hospital Pulido Valente, Lisbon
  - Hospital São João, Porto
- Institutul de Pneumoftiziologie "Marius Nasta", Bucharest, Romania
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital - Yonsei University Health System - Pulmonary, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Hospital Universitario de Bellvitge, Barcelona, Catalonia, Spain
- Turkey (Türkiye) (3):
  - Ege University Hospital - Department of Pulmonology, Bornova, İzmir
  - Health Sciences University Gulhane Training and Research Hospital, Ankara
  - Yedikule Chest Disease and Surgery Training and Research Hospital, Istanbul
- Royal Brompton and Harefield NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trapnell BC, Inoue Y, Bonella F, Wang T, McCarthy C, Arai T, Akasaka K, Mariani F, Mogulkoc N, Song JW, Baba T, Jouneau S, Numakura T, Ocal N, Mihaltan F, Ataya A, Bendstrup E, Campo I, Carey B, Arena R, Robinson B, Fleming R, Wasfi Y, Pratt R; IMPALA-2 Trial Investigators. Phase 3 Trial of Inhaled Molgramostim in Autoimmune Pulmonary Alveolar Proteinosis. N Engl J Med. 2025 Aug 21;393(8):764-773. doi: 10.1056/NEJMoa2410542. PMID 40834301

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatient Medical Clinics 19 May 2021 -16 June 2023
Pre-assignment Details: Two screening visits were conducted 6 and 3 weeks prior to the Day 1 baseline visit. At the baseline visit, eligible subjects were centrally randomized through a Randomization and Trial Supply Management system to 48 weeks of double-blind treatment with MOL-OD or PBO.
  To be randomized patients were required to have a percent predicted DLCO adjusted for hemoglobin (%DLCOadj) of 70% or less and no variation in %DLCOadj of +/-15%.
Groups:
- Molgramostim: Double-blind treatment with molgramostim nebulizer solution 300 µg once daily for 48 weeks
  Molgramostim: Molgramostim 300 µg nebulizer solution
- Placebo: Double-blind treatment with placebo nebulizer solution once daily for 48 weeks
  Placebo: Matching placebo nebulizer solution
Period: Double-blind
Arm/Group | Molgramostim | Placebo
Started | 81 | 83
Completed | 79 | 80 (one subject in Placebo discontinued blinded IMP but completed all study visits and assessments)
Not Completed | 2 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Open-Label Extension
Arm/Group | Molgramostim | Placebo
Started | 79 | 81 (One subject discontinued IMP in the double-blind period and completed all study visits then entered the OLE)
Completed | 0 | 0
Not Completed | 79 | 81
Not completed — Study ongoing | 79 | 81

BASELINE CHARACTERISTICS:
Population: One subject in the placebo group stopped randomized drug but continued in the study to complete all visits and assessments
Groups:
- Total: Total of all reporting groups
Arm/Group | Molgramostim | Placebo | Total
Number analyzed (Participants) | 81 | 83 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (13.03) | 48.4 (12.69) | 49.6 (12.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 29 | 66
  Male | 44 | 54 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 36 | 37 | 73
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 38 | 40 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  Romania | 4 | 2 | 6
  United States | 11 | 12 | 23
  Japan | 29 | 24 | 53
  United Kingdom | 1 | 2 | 3
  Portugal | 0 | 1 | 1
  Spain | 2 | 0 | 2
  Canada | 5 | 2 | 7
  South Korea | 6 | 10 | 16
  Turkey | 8 | 10 | 18
  Belgium | 0 | 1 | 1
  Ireland | 2 | 0 | 2
  Poland | 0 | 3 | 3
  Italy | 4 | 5 | 9
  Australia | 0 | 1 | 1
  France | 5 | 4 | 9
  Germany | 4 | 6 | 10
%DLCOadj at Baseline [Median (Full Range); unit: %] — Percent predicted diffusion capacity for carbon monoxide adjusted for hemoglobin concentration.
  % | 54.0 [25 to 72] | 55.0 [28 to 71] | 55 [25 to 72]
%DLCOadj at Randomization <=50% [Count of Participants; unit: Participants] — Percent predicted diffusion capacity for carbon monoxide adjusted for hemoglobin concentration less than or equal to 50% predicted.
  Participants | 31 | 32 | 63
%DLCOadj at Randomization >50% [Count of Participants; unit: Participants] — Percent predicted diffusion capacity for carbon monoxide adjusted for hemoglobin concentration greater than 50%
  Participants | 50 | 51 | 101

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Percent (%) Predicted Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) Adjusted for Hemoglobin Concentration to Week 24
Description: As a measure of pulmonary gas transfer, a standardized lung function test, DLCO, was conducted. The single-breath DLCO test was performed in accordance with American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines for DLCO testing. Results reported as % predicted DLCO adjusted for hemoglobin concentration (%predicted DLCOadj).
Time Frame: From Baseline to Week 24
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: % predicted DLCO adjusted for hemoglobin
Arm/Group | Molgramostim | Placebo
Number analyzed (Participants) | 81 | 83
% predicted DLCO adjusted for hemoglobin | 9.8 [7.3 to 12.3] | 3.8 [1.4 to 6.3]
Statistical Analysis 1: Comparison: Molgramostim vs Placebo; Test type: Superiority; p = 0.0007, Mixed Models Analysis; Modelled using MMRM adjusted for baseline % predicted DLCOadj, treatment, visit, region, severity stratification and treatment-visit interaction; Mean Difference (Net) = 6.0, 95% CI 2-sided [2.5 to 9.4] — Difference from placebo

2. Secondary Outcome: Change From Baseline in Percent (%) Predicted DLCO Adjusted for Hemoglobin Concentration (%DLCOadj) to Week 48
Description: As a measure of pulmonary gas transfer, a standardized lung function test, DLCO, was conducted. The single-breath DLCO test was performed in accordance with American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines for DLCO testing. Results reported as % predicted DLCO adjusted for hemoglobin concentration (%predicted DLCOadj). Higher values indicate better respiratory gas exchange.
Time Frame: From Baseline to Week 48
Measure: Least Squares Mean (95% Confidence Interval); unit: Unit of Measure: % predicted DLCO adjust
Arm/Group | Molgramostim | Placebo
Number analyzed (Participants) | 81 | 83
Unit of Measure: % predicted DLCO adjust | 11.6 [8.7 to 14.5] | 4.7 [1.8 to 7.6]
Statistical Analysis 1: Comparison: Molgramostim vs Placebo; Test type: Superiority; p = 0.0008, Mixed Models Analysis — Modelled using MMRM adjusted for baseline % predicted DLCOadj, treatment, visit, region, severity stratification and treatment-visit interaction; Mean Difference (Net) = 6.9, 95% CI 2-sided [2.9 to 10.9] — Difference from Placebo

3. Secondary Outcome: Change From Baseline in St. Georges Respiratory Questionnaire (SGRQ) Total Score to Week 24
Description: The Saint Georges Respiratory Questionnaire (SGRQ) is designed to measure respiratory health impairment. The scale includes questions related to three components: Activity (activities that cause or are limited by breathlessness), Impact (social functioning and psychological disturbances resulting from airway disease), and Symptoms (respiratory symptoms, their frequency and severity). The questionnaire has a recall period of 4 weeks for Symptoms, whereas Activity and Impact components address the subject's current state. SGRQ scored on a 0-100 scale with lower scores indicating better respiratory health.
Time Frame: From Baseline to Week 24
Measure: Least Squares Mean (95% Confidence Interval); unit: Change from baseline units on a scale
Arm/Group | Molgramostim | Placebo
Number analyzed (Participants) | 81 | 83
Change from baseline units on a scale | -11.5 [-15.01 to -7.98] | -4.9 [-8.28 to -1.52]
Statistical Analysis 1: Comparison: Molgramostim vs Placebo; Test type: Superiority; p = 0.0072, Mixed Models Analysis; Mean Difference (Net) = -6.59, 95% CI 2-sided [-11.40 to -1.79]

4. Secondary Outcome: Change From Baseline in SGRQ Activity Component Score to Week 24
Description: The Saint Georges Respiratory Questionnaire (SGRQ) Activity scale is a subscale of the SGRQ and is designed to measure the effect of respiratory health impairment on daily activity affected by breathlessness. The questionnaire for the Activity components addresses the subject's current state. SGRQ Activity is scored on a 0-100 scale with lower scores indicating better respiratory health activity
Time Frame: From Baseline to Week 24
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Molgramostim | Placebo
Number analyzed (Participants) | 81 | 83
units on a scale | -13.03 [-17.58 to -8.49] | -5.22 [-9.76 to -0.69]
Statistical Analysis 1: Comparison: Molgramostim vs Placebo; Test type: Superiority; p = 0.0149, Mixed Models Analysis; Mean Difference (Net) = -7.81, 95% CI 2-sided [-14.10 to -1.52]

5. Secondary Outcome: Change From Baseline in Exercise Capacity (EC), Expressed as Peak Metabolic Equivalents (METs) to Week 24
Description: As a functional measure of exertional limitations related to dyspnea, EC was assessed by an exercise treadmill test. EC was expressed in peak METs (1 MET=3.5 mL O2/kg/min). The highest treadmill speed and grade achieved was used to calculate peak METs. Higher values indicate better functional capacity.
Time Frame: From Baseline to Week 24
Measure: Least Squares Mean (95% Confidence Interval); unit: Change from baseline in METS
Arm/Group | Molgramostim | Placebo
Number analyzed (Participants) | 81 | 83
Change from baseline in METS | 1.11 [0.76 to 1.46] | 0.70 [0.34 to 1.05]
Statistical Analysis 1: Comparison: Molgramostim vs Placebo; Test type: Superiority; p = 0.0845, Mixed Models Analysis; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [-0.06 to 0.89]

6. Secondary Outcome: Change From Baseline in SGRQ Total Score to Week 48
Description: as for outcome 3
Time Frame: From Baseline to Week 48
Measure: Least Squares Mean (95% Confidence Interval); unit: Change from baseline units on a scale
Arm/Group | Molgramostim | Placebo
Number analyzed (Participants) | 81 | 83
Change from baseline units on a scale | -10.72 [-15.01 to -6.44] | -5.85 [-9.96 to -1.74]
Statistical Analysis 1: Comparison: Molgramostim vs Placebo; Test type: Superiority; p = 0.1046, Mixed Models Analysis; Mean Difference (Net) = -4.87, 95% CI 2-sided [-10.76 to 1.01]

7. Secondary Outcome: Change From Baseline in SGRQ Activity From Baseline to Week 48
Description: as for outcome 4
Time Frame: From Baseline to Week 48
Measure: Least Squares Mean (95% Confidence Interval); unit: Change from baseline score on a scale
Arm/Group | Molgramostim | Placebo
Number analyzed (Participants) | 81 | 83
Change from baseline score on a scale | -13.39 [-18.87 to -7.91] | -7.40 [-12.72 to -2.09]
Statistical Analysis 1: Comparison: Molgramostim vs Placebo; Test type: Superiority; p = 0.1216, Mixed Models Analysis; Mean Difference (Net) = -5.99, 95% CI 2-sided [-13.57 to 1.59]

8. Secondary Outcome: Change From Baseline in EC, Expressed as Peak METs to Week 48
Description: as for outcome 5
Time Frame: From Baseline to Week 48
Measure: Least Squares Mean (95% Confidence Interval); unit: Change from baseline in METS
Arm/Group | Molgramostim | Placebo
Number analyzed (Participants) | 81 | 83
Change from baseline in METS | 1.13 [0.77 to 1.49] | 0.58 [0.22 to 0.93]
Statistical Analysis 1: Comparison: Molgramostim vs Placebo; Test type: Superiority; p = 0.0234, Mixed Models Analysis; Mean Difference (Final Values) = 0.55, 95% CI 2-sided [0.07 to 1.03] — Change from baseline compared to placebo

9. Secondary Outcome: Change From Baseline in Alveolar-arterial Oxygen Difference (A-aDO2) to Week 24 (All Subjects)
Description: A-aDO2 was used as an additional measure of gas exchange.
Time Frame: From Baseline to Week 24
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Molgramostim | Placebo
Number analyzed (Participants) | 81 | 83
mmHg | -7.97 [-11.62 to -4.32] | -3.96 [-7.48 to -0.44]
Statistical Analysis 1: Comparison: Molgramostim vs Placebo; Test type: Superiority; p = 0.1043, Mixed Models Analysis; Mean Difference (Final Values) = -4.01, 95% CI 2-sided [-8.84 to 0.83]

10. Secondary Outcome: Number of Subjects With Serious and Non-serious Adverse Events
Description: Assessment of the safety of molgramostim compared to placebo
Time Frame: From Baseline until End of Double-blind treatment (Week 48)
Measure: Number; unit: participants
Arm/Group | Molgramostim | Placebo
Number analyzed (Participants) | 81 | 83
participants
  Any TEAE | 69 | 71
  Any TESAE | 14 | 20

11. Secondary Outcome: Number of Subjects With Positive Treatment-boosted Anti Granulocyte Macrophage Colony Stimulating Factor (GM-CSF) Antibody Titers During 24 Weeks' Treatment and During 48 Weeks' Treatment
Description: Assess the effect of molgramostim or placebo on antiGM-CSF antibody titers that increased by a dilution factor of 2.(4X increase in titer compared to Baseline).
Time Frame: From Baseline until End of Double-blind treatment Week-48
Population: One subject in the molgramostim group had missing antiGM-CSF titers.
Measure: Count of Participants; unit: Participants
Arm/Group | Molgramostim | Placebo
Number analyzed (Participants) | 81 | 83
Participants
  Week 24: number analyzed (Participants) | 80 | 83
  Week 24 | 28 | 30
  Week 48: number analyzed (Participants) | 80 | 83
  Week 48 | 39 | 37

12. Secondary Outcome: Changes in Forced Vital Capacity (FVC) %Predicted Normal
Description: Forced vital capacity is the volume of air that can be expired after a deep breath. Higher volumes indicate better respiratory function. FVC is scored as % of predicted normal expired vital capacity.
Time Frame: From Baseline to Weeks 24 and 48
Measure: Mean (Standard Deviation); unit: % FVC predicted
Arm/Group | Molgramostim | Placebo
Number analyzed (Participants) | 78 | 81
% FVC predicted
  Week 24 | 3.2 (6.20) | 0.9 (5.74)
  Week 48 | 3.2 (7.92) | -0.1 (8.27)

13. Secondary Outcome: Changes in Forced Expiratory Volume in One Second (FEV1) % Predicted Normal.
Description: FEV1 is the volume of air expired in 1 second in liters (L). Higher values indicate better respiratory function.
Time Frame: From Baseline to Weeks 24 and 48
Measure: Mean (Standard Deviation); unit: %predicted normal
Arm/Group | Molgramostim | Placebo
Number analyzed (Participants) | 78 | 81
%predicted normal
  Week 24 | 1.2 (7.08) | -0.3 (5.35)
  Week 48 | 1.4 (7.98) | -1.4 (7.56)

14. Secondary Outcome: Change in QT Interval Corrected by Fridericia (QTcF)
Description: Assessment of the safety of MOL compared to placebo
Time Frame: From Baseline to Weeks 4 and 24
Population: Some subjects did not have ECG obtained at some visits.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Molgramostim | Placebo
Number analyzed (Participants) | 81 | 83
msec
  Week 4: number analyzed (Participants) | 80 | 83
  Week 4 | -2.51 (10.543) | 1.59 (10.127)
  Week 24: number analyzed (Participants) | 79 | 80
  Week 24 | -1.89 (13.190) | -0.96 (11.534)

ADVERSE EVENTS:
Time Frame: Adverse events during double-blind treatment (48 Weeks)
Description: Adverse events only reported for the 48-week double-blind part of the study. The open label extension is currently ongoing and has not been analyzed. Results will be reported when the open-label study is complete.
Groups:
- Molgramostim: Double-blind treatment with molgramostim nebulizer solution 300 µg once daily for 48 weeks
  Molgramostim: Molgramostim 300 µg nebulizer solution
  79 subjects completed double-blind treatment and continued in the open-label extension. The open-label study is still ongoing.
- Placebo: Double-blind treatment with placebo nebulizer solution once daily for 48 weeks
  Placebo: Matching placebo nebulizer solution
  81 subjects completed double-blind treatment and enrolled in the open-label extension. The open-label study is still ongoing.
Arm/Group | Molgramostim | Placebo
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/83
Serious Adverse Events (participants affected / at risk) | 14/81 | 20/83
Other Adverse Events (participants affected / at risk) | 69/81 | 71/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Molgramostim (N=81) | Placebo (N=83)
Alveolar proteinosis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 9 (9) — Worsening of aPAP
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Mycobacterium avium complex infection (Infections and infestations) | 1 (1) | 0 (0)
Brain abscess (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Delusion (Psychiatric disorders) | 1 (1) | 0
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Intracranial mass (Nervous system disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Molgramostim (N=81) | Placebo (N=83)
Covid-19 (Infections and infestations) | 16 (17) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (30) | 18 (23)
Nasopharyngitis (Infections and infestations) | 11 (19) | 7 (9)
Pyrexia (General disorders) | 11 (16) | 9 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 9 (10) | 2 (3)
Headache (Nervous system disorders) | 9 (33) | 7 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3)
Dizziness (Nervous system disorders) | 7 (8) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (5)
Non-cardiac chest pain (General disorders) | 7 (8) | 5 (8)
Nausea (Gastrointestinal disorders) | 6 (10) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (12) | 3 (3)
Vomiting (Gastrointestinal disorders) | 6 (7) | 1 (1)
Bronchitis (Infections and infestations) | 5 (5) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 1 (2)
Alveolar proteinosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) — Worsening of aPAP
Hypertension (Vascular disorders) | 4 (5) | 5 (5)
Fatigue (General disorders) | 2 (2) | 6 (8)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 3 (4)
Urinary tract infection (Infections and infestations) | 4 (4) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT04544293/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-24): https://cdn.clinicaltrials.gov/large-docs/93/NCT04544293/SAP_001.pdf